CLINICAL TRIAL: NCT05257954
Title: Frailty in Patient Undergoing Percutaneous Left Atrial Appendage Closure The Frail-LAAC Study
Brief Title: Frailty in Patient Undergoing Percutaneous Left Atrial Appendage Closure.
Acronym: Frail-LAAC
Status: Recruiting | Type: Observational
Sponsor: Josep Rodes-Cabau (Other)
Responsible Party: Sponsor-Investigator, Josep Rodes-Cabau, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: Frail-LAAC
Record Dates: First submitted 2022-02-10; First posted 2022-02-25 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Transcatheter Left Atrial Appendage Closure; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prevalence and severity of frailty in patients undergoing LAAC, as well as its association to peri-procedural and long-term outcomes and quality of life.

DETAILED DESCRIPTION:
Transcatheter left atrial appendage closure (LAAC) has emerged as an alternative to anticoagulation for preventing thromboembolic events in patients with non-valvular atrial fibrillation and relative or absolute contraindications to oral anticoagulation (OAC).

Procedural safety and success are now excellent with approximately 98% of successful procedures without major complications. LAAC seems to offer persisting protection against ischemic events in long-term reports, while also decreasing bleeding risk by reducing antithrombotic treatment intensity. However, patients undergoing LAAC in real-world practice are a high-risk population with a high rate of adverse events, mainly not related to the LAAC device-procedure. As a prophylactic intervention, the beneficial effects of LAAC increase over time, as more potential adverse events (ischemic and haemorrhagic) are prevented. Thus, it took approximately 5 years to reach cost-effectiveness (favoring LAAC versus oral anticoagulation) in the pooled data from PROTECT-AF and PREVAIL randomized controlled trials. Patients that experience early death after LAAC do not fully benefit from the costly procedure - that can be therefore considered futile. In a recent study, close to 1 on 5 LAAC recipient had either died or suffered from a major ischemic event within the first year after the procedure highlighting the need for better patient selection before LAAC.

The definition of frailty is nonconsensual and has constantly evolved in the literature. Nonetheless, there is a general agreement that frailty is a multidimensional concept involving many domains (such as nutrition, mobility, strength and cognitive) and that frail patients are a high-risk population and vulnerable to stressors and adverse outcomes. Thus, considering this global definition, assessing frailty using multidomain scales is more appropriate to discriminate frail to non-frail patients.

Frailty and its association to adverse events are well-known in transcatheter aortic valve replacement (TAVR). Despite being performed in a high-risk population, frailty has not yet been studied in LAAC although it could be a potent indicator for futile or harmful procedures. The implementation of frailty assessment into the routine practice could help identify vulnerable patients who will most likely less benefit from the LAAC procedure. Therefore, in this prospective multicenter trial, the investigators seek to explore frailty and its consequences in LAAC recipients.

ELIGIBILITY:
Inclusion Criteria:

* Transcatheter LAAC with any approved device
* Age ≥18 years old

Exclusion Criteria:

* Unable to provide informed consent
* Severe neuropsychiatric impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old undergoing Transcatheter LAAC with any approved device
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of frailty | Baseline (before transcatheter Left Atrial Appendage Closure)
  Evaluated with Clinical Frailty Scale (CFS) 9-point scale (1-Very fit to 9-Terminally ill)
Prevalence of frailty | Baseline (before transcatheter Left Atrial Appendage Closure)
  Evaluated with Essential Frailty Toolset (EFT) (Scored 0 (least frail) to 5 (most frail)
Rate of all-cause mortality | 1-year follow-up
Rate of ischemic events | 1-year follow-up
  Stroke
Rate of all-cause mortality and ischemic events | 1-year follow-up
  all-cause mortality and Stroke

SECONDARY OUTCOMES:
Rate of All-cause mortality | 2, 3, 4 and 5-year follow-up
Rate of ischemic events | 2, 3, 4 and 5-year follow-up
  Ischemic stroke or peripheral embolism
Rate of all-cause mortality and ischemic events | 2-, 3-, 4- and 5-year follow-up
  Rate of death from any cause + ischemic stroke or peripheral embolism
Rate of Rehospitalisation | 1-, 2-, 3-, 4- and 5-year follow-up
  Rate of any readmission to a hospital
Number of participants discharged to a healthcare facility | 1-month follow-up
  Number of participants discharged to convalescence center, rehabilitation center, assisted-living center, or nursing home; excluding those previously living in a facility.
Rate of bleeding | 1-, 2-, 3-, 4- and 5-year follow-up
  Minor, Major and Life-threatening Bleeding
Changes in quality of life | Baseline (before transcatheter Left Atrial Appendage Closure) and 1-year follow-up
  Evaluated with EQ5-D questionnaire (5 dimensions questionnaire: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels : no problems, slight problems, moderate problems, severe problems and extreme problems.)

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ_UL, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asmarats L, Rodes-Cabau J. Percutaneous Left Atrial Appendage Closure: Current Devices and Clinical Outcomes. Circ Cardiovasc Interv. 2017 Nov;10(11):e005359. doi: 10.1161/CIRCINTERVENTIONS.117.005359. PMID 29146668
- [Result] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Result] Landmesser U, Tondo C, Camm J, Diener HC, Paul V, Schmidt B, Settergren M, Teiger E, Nielsen-Kudsk JE, Hildick-Smith D. Left atrial appendage occlusion with the AMPLATZER Amulet device: one-year follow-up from the prospective global Amulet observational registry. EuroIntervention. 2018 Aug 3;14(5):e590-e597. doi: 10.4244/EIJ-D-18-00344. PMID 29806820
- [Result] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Result] Holmes DR Jr, Reddy VY, Gordon NT, Delurgio D, Doshi SK, Desai AJ, Stone JE Jr, Kar S. Long-Term Safety and Efficacy in Continued Access Left Atrial Appendage Closure Registries. J Am Coll Cardiol. 2019 Dec 10;74(23):2878-2889. doi: 10.1016/j.jacc.2019.09.064. PMID 31806131
- [Result] Mesnier J, Cruz-Gonzalez I, Peral V, Nombela-Franco L, Freixa X, Laffond AE, Mas-Llado C, McInerney A, Regueiro A, O'Hara G, Rodes-Cabau J. Ten-Year Outcomes Following Percutaneous Left Atrial Appendage Closure in Patients With Atrial Fibrillation and Absolute or Relative Contraindications to Chronic Anticoagulation. Circ Cardiovasc Interv. 2021 Aug;14(8):e010821. doi: 10.1161/CIRCINTERVENTIONS.121.010821. Epub 2021 Jul 16. No abstract available. PMID 34266312
- [Result] Panikker S, Lord J, Jarman JW, Armstrong S, Jones DG, Haldar S, Butcher C, Khan H, Mantziari L, Nicol E, Hussain W, Clague JR, Foran JP, Markides V, Wong T. Outcomes and costs of left atrial appendage closure from randomized controlled trial and real-world experience relative to oral anticoagulation. Eur Heart J. 2016 Dec 7;37(46):3470-3482. doi: 10.1093/eurheartj/ehw048. Epub 2016 Mar 1. PMID 26935273
- [Result] Hoogendijk EO, Afilalo J, Ensrud KE, Kowal P, Onder G, Fried LP. Frailty: implications for clinical practice and public health. Lancet. 2019 Oct 12;394(10206):1365-1375. doi: 10.1016/S0140-6736(19)31786-6. PMID 31609228
- [Result] Dent E, Kowal P, Hoogendijk EO. Frailty measurement in research and clinical practice: A review. Eur J Intern Med. 2016 Jun;31:3-10. doi: 10.1016/j.ejim.2016.03.007. Epub 2016 Mar 31. PMID 27039014
- [Result] Kim DH, Kim CA, Placide S, Lipsitz LA, Marcantonio ER. Preoperative Frailty Assessment and Outcomes at 6 Months or Later in Older Adults Undergoing Cardiac Surgical Procedures: A Systematic Review. Ann Intern Med. 2016 Nov 1;165(9):650-660. doi: 10.7326/M16-0652. Epub 2016 Aug 23. PMID 27548070
- [Result] Rodriguez-Manas L, Feart C, Mann G, Vina J, Chatterji S, Chodzko-Zajko W, Gonzalez-Colaco Harmand M, Bergman H, Carcaillon L, Nicholson C, Scuteri A, Sinclair A, Pelaez M, Van der Cammen T, Beland F, Bickenbach J, Delamarche P, Ferrucci L, Fried LP, Gutierrez-Robledo LM, Rockwood K, Rodriguez Artalejo F, Serviddio G, Vega E; FOD-CC group (Appendix 1). Searching for an operational definition of frailty: a Delphi method based consensus statement: the frailty operative definition-consensus conference project. J Gerontol A Biol Sci Med Sci. 2013 Jan;68(1):62-7. doi: 10.1093/gerona/gls119. Epub 2012 Apr 16. PMID 22511289
- [Result] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Result] Hinterbuchner L, Strohmer B, Hammerer M, Prinz E, Hoppe UC, Schernthaner C. Frailty scoring in transcatheter aortic valve replacement patients. Eur J Cardiovasc Nurs. 2016 Oct;15(6):384-97. doi: 10.1177/1474515115596640. Epub 2015 Jul 27. PMID 26216870
- [Result] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869